CLINICAL TRIAL: NCT02984592
Title: Regular Physical Activity Improves Ejaculation Time and Patient-reported Outcomes
Brief Title: Effect of Exercise on Premature Ejaculation
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, M.D., Ankara Training and Research Hospital
Other Study IDs: 5006
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation; intravaginal ejaculatory latency time; premature ejaculation diagnostic tools
MeSH Terms: conditions — Premature Ejaculation | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: The participants in group 1 will state that they participate regular exercise programs in the previous 6 months
  Interventions: Behavioral: physical exercise
- Group 2: The participants in group 2 will state that they do not perform any regular exercise in previous 6 months.

INTERVENTIONS:
Behavioral: physical exercise — regular exercise programs in the previous 6 months.
  Groups: Group 1

SUMMARY:
Premature ejaculation (PE) is one of the prevalent disorders in men; its leading sequel such as lack of self-confidence, anxiety, depression and unsatisfactory intercourse in men and their partners. The current study was aimed to evaluate the relationship between ejaculation and physical activity.

DETAILED DESCRIPTION:
Premature ejaculation (PE) is the most frequent sexual dysfunction in males, and its prevalence has been reported as 21-33%. Currently, there are no universal criteria for the diagnosis, or treatment strategies or approaches for PE. Lack of observational studies directed to PE makes comprehension of this sexual dysfunction difficult. The common point for definition of PE is a short duration between penetration and ejaculation, little or no control on voluntary control of ejaculation, and annoying character and negative effect of this condition on the individual. There are various treatment methods since ejaculation physiology and neuroanatomy is not yet clearly demonstrated. According to neurobiological hypothesis of Waldinger, a dysfunction in the serotonin pathway of the central system such as serotonin-2C hyposensitivity and/or serotonin-1A receptor hypersensitivity is a possible cause of lifelong PE. These experimental animal models showed that serotonergic activity at hypothalamic level inhibited ejaculation reflex. Based on this physiological effect, selective serotonin reuptake inhibitors (SSRI), and serotonin agonists increase intravaginal ejaculation latency time (IELT). A number of studies showed that exercise increased the functional effect of serotonin in the human brain.

The effects of physical activity level on human health have attracted interest worldwide. Lack of physical activity forms the basis of various health problems, however regular physical act contributes prevention and treatment of a number of disorders.

In current study, investigators will compare the ejaculation control, IELT, and prevalence of PE between sportsmen that have regular physical activity, and the individuals with a sedentary lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* 18-45-year-old
* sexually active
* heterosexual,without erectile dysfunction
* sexual partner for at least six months, and sexual intercourse at least twice a week

Exclusion Criteria:

* chronic systemic disorders (such as diabetes or hypertension)
* use of narcotic/hypnotic drugs or stimulants
* anabolic steroids
* selective serotonin receptors inhibitors
* previous diagnosis and treatment for PE

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants are 18-45 year-old, and have regular sexual activity for at least 6 months. A comparison was made by metabolic equivalents (MET), premature ejaculation diagnostic tool (PEDT) and intravaginal ejaculatory latency time (IELT).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
intravaginal ejaculatory latency time | 1 month
  IELT value (second) according to the duration determined by the sexual partner with stopwatch method

SECONDARY OUTCOMES:
Premature ejaculation diagnostic tool score | 1 month
  Premature Ejaculation Diagnostic Tool (PEDT) includes five items; control, frequency, minimal stimulation, distress, and interpersonal difficulty. In this classification tool, score 8 indicates no premature ejaculation, scores 9 and 10 indicate possible premature ejaculation, and scores equal or higher than 11 indicates premature ejaculation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pastore AL, Palleschi G, Leto A, Pacini L, Iori F, Leonardo C, Carbone A. A prospective randomized study to compare pelvic floor rehabilitation and dapoxetine for treatment of lifelong premature ejaculation. Int J Androl. 2012 Aug;35(4):528-33. doi: 10.1111/j.1365-2605.2011.01243.x. Epub 2012 Feb 9. PMID 22320846
- [Result] Pastore AL, Palleschi G, Fuschi A, Maggioni C, Rago R, Zucchi A, Costantini E, Carbone A. Pelvic floor muscle rehabilitation for patients with lifelong premature ejaculation: a novel therapeutic approach. Ther Adv Urol. 2014 Jun;6(3):83-8. doi: 10.1177/1756287214523329. PMID 24883105